CLINICAL TRIAL: NCT04985006
Title: Effect of Exercise Intensity on Epigenetic Response in Healthy Young Adult
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rahmaningsih Mara Sabirin (Other)
Collaborators: Indonesia Endowment Fund for Education (LPDP), Ministry of Finance Republik of Indonesia (Unknown)
Responsible Party: Sponsor-Investigator, Rahmaningsih Mara Sabirin, Principal investigator, Doctoral students, Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: RMS01
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: microRNA; exercise; aerobic exercise; epigenetic; mitochondrial biogenesis
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: All the participant will be asked to run in moderate and high intensity in random order. The interval between the first exercise and the next is 48 hours to 14 days.
Who Masked: Outcomes Assessor
Masking Description: The outcome measurement (microRNA measurement using qPCR and PGC 1 alpha measurement using ELISA) will be done by professional laboratory assistant who is blind about the intervention given to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity aerobic exercise (Experimental): each subject will undergo running in medium intensity.
  Interventions: Behavioral: running at moderate intensity
- High intensity aerobic exercise (Active Comparator): each subject will undergo running in high intensity.
  Interventions: Behavioral: running at high intensity

INTERVENTIONS:
Behavioral: running at moderate intensity — intensity was determined by calculating the subject's heart rate reserve using the formula: ((resting heart rate maximal - resting heart rate) x % of target intensity) + resting heart rate. At moderate intensity, the subject will be asked to run at 50-59% Heart rate reserve (HRR) for 30 minutes from the time the target intensity is reached.
  Arms: Moderate intensity aerobic exercise
Behavioral: running at high intensity — intensity was determined by calculating the subject's heart rate reserve using the formula: ((resting heart rate maximal - resting heart rate) x % of target intensity) + resting heart rate. At moderate intensity, the subject will be asked to run at 70-75% HRR for 30 minutes from the time the target intensity is reached.
  Arms: High intensity aerobic exercise

SUMMARY:
Aerobic exercise has been shown to trigger a variety of body responses which then trigger physiological adaptations. One of the physiological adaptations that occur is an increase in mitochondrial biogenesis. Mitochondria are organelles in cells that play a role in providing energy. An increase in the number of mitochondria will increase the supply of energy for muscle cell contraction, so that muscles do not get tired easily.

Mitochondrial biogenesis is known to be regulated by Peroxisome proliferator-activated receptor gamma co-activator-1 alpha (PGC-1α), by inducing transcription of genes encoded by the nucleus and mitochondria. Peroxisome proliferator-activated receptor gamma co-activator-1 alpha is a protein which encoded by the PPARGC1A gene. PPARGC1A gene expression itself can be influenced by microRNA, a short non-coding RNA that can regulate gene expression by suppressing or degrading the target gene. In vitro studies show that PPARGC1A gene is a direct gene target of microRNA (miR)-23a.

In human studies, aerobic exercise has been shown to reduce miR-23a levels in human muscles immediately after exercise. Another study found an increase in muscle PGC-1 alpha levels after exercise. In addition to being detectable in muscle, both miR-23a and PGC-1 alpha can be measured in blood plasma. However, whether exercise can reduce miR-23a levels while increasing PGC-1 alpha levels in circulation, still needs further research. Therefore, this study aims to examine whether aerobic exercise will reduce miR-23a levels and PGC-1 alpha levels in plasma. In addition, this study will also compare whether exercise intensity affects the expression of miR-23a and PGC-1 alpha.

In this study, measurements will be made on blood plasma to reduce the level of invasiveness. Subjects will be asked to come to the laboratory three times. The first meeting consisted of an examination, while in the second and third meetings the subjects would be asked to run at a moderate or high intensity. Blood sampling will be done before and after exercise.

DETAILED DESCRIPTION:
This study is a randomized cross-over trial with a pre and post intervention measurement. In general, each subject will be asked to run with moderate and vigorous intensity in a random order. Healthy males aged 18-25 were recruited through announcements on social media. Subjects who are willing to join are asked to fill out a form via google forms. Subjects who meet the inclusion and exclusion criteria will be asked to come to the laboratory. At the first meeting, participants will be examined to ensure the subject meets the criteria. The examinations conducted including measurement of body weight, body height, blood pressure, lung function, and electrocardiography. Body weight will be measured using a digital weight scale, while body height will be measured three times using a stadiometer. For measuring the a blood pressure, the subject was asked to lie down for at least 5 minutes. Blood pressure will be measured three times on the right arm using the Omron digital sphygmomanometer. Lung function examination including forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and maximal voluntary ventilation (MVV) will be measured using a spirometer. Following the standard procedure from American Thoracic Society/ European Respiratory Society regarding spirometry examination, measurements will be performed in an upright sitting position. Measurement of FVC and FEV1 will be performed at least three times, while MVV will be performed at least twice to obtain reliable and acceptable results. Only healthy subject will be included in the study.

At least 48 hours to 14 days after the first meeting, subjects will be asked to come to the second and third meetings to do moderate or high intensity exercise in randomized order. Before and after exercise, 3 ml of blood will be drawn from the cubital vein and put in an Ethylenediamine tetra acetic acid (EDTA) tube to collect the plasma. The plasma will then be centrifuged to separate the plasma from the blood cells. Plasma is stored in the freezer -80 degrees celsius until it will be used.

The microRNA levels before and after exercise will be measured using real time polymerase chain reaction (qPCR). In general, RNA extraction will be conduct using the plasma extraction kit, following by complement DNA synthesis and qPCR. Normalization will be conduct by adding 3.5 micro liters of cel-miR-39 spike in control to each sample. Quantification of the microRNA level will be expressed as 2-[(CT microRNA)-(CT cel-miR-39)].

Normality test will be performed using Shapiro-Wilk test. If the data is normally distributed, the statistical test of the measurement results before and after exercise at both intensities will be analyzed using independent t-test. Meanwhile, if the data is not normally distributed, statistical analysis will be done using Mann Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI <30
* systolic blood pressure <140 mmHg
* diastolic blood pressure <90 mmHg
* have no chronic disease
* have no complaints related to the musculoskeletal, respiratory and cardiovascular systems
* willing to to come to the laboratory
* willing to sign the informed consent form

Exclusion Criteria:

* suffer from chronic disease
* have complaints related to the musculoskeletal, respiratory, and cardiovascular systems
* have a history of smoking, both active and passive in the past year

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
miR-23a level in plasma | Before and immediately after exercise
  microRNA level will be measured using qpCR. Ce-miR-39 spike in control will be added for normalization. Quantification of the microRNA level will be expressed as 2-[(CT microRNA)-(CT cel-miR-39)].
PGC 1 alpha level in plasma | Before and immediately after exercise
  PGC 1 alpha level will be measured using ELISA. The result will be obtained in nanograms.

CONTACTS AND LOCATIONS:
Overall Officials: Rahmaningsih M Sabirin, MD, M.Sc, Principal Investigator — Department of Physiology. Faculty of Medicine, Public Health and Nursing. Universitas Gadjah Mada
Locations (1):
- Department of Physiology. Faculty of Medicine, Public Health and Nursing, Universitas Gadjah Mada, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No